CLINICAL TRIAL: NCT05309525
Title: Effect of Oral TXA on Buttock Bruising Post CCH Injections in Adult Females
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Luxurgery (Industry)
Responsible Party: Principal Investigator, Sachin Shridharani, Medical Director, LUXURGERY, Luxurgery
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: LUX-EN-001
Record Dates: First submitted 2022-03-24; First posted 2022-04-04 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2023-03

CONDITIONS: Cellulite
MeSH Terms: conditions — Cellulite | interventions — Tranexamic Acid; Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Cohort A (Active Comparator): Per treatment area, subjects will be injected with up to 0.84 mg of QWO as 12 subcutaneous injections (0.3-mL injection administered as three 0.1-mL aliquots per injection), dependent on the amount of dimples (0.3 ml per dimple). A treatment area is defined as a left or right buttock, so patients may receive up to 1.84 mg, or 24 injections total (2 areas per treatment visit). The minimum dosage of QWO will be 0.92 mg, or 6 injections per treatment area (2 areas per treatment visit.
  Cohort A subjects will be given 1300 mg tranexamic acid PO TID prior to the day of the first CCH injections, the day of the first CCH injections, and the 3 days following the first CCH injections.
  Interventions: Drug: Collagenase Clostridium Histolyticum-Aaes; Drug: Lysteda 650 MG Oral Tablet
- Cohort B (Active Comparator): Per treatment area, subjects will be injected with up to 0.84 mg of QWO as 12 subcutaneous injections (0.3-mL injection administered as three 0.1-mL aliquots per injection), dependent on the amount of dimples (0.3 ml per dimple). A treatment area is defined as a left or right buttock, so patients may receive up to 1.84 mg, or 24 injections total (2 areas per treatment visit). The minimum dosage of QWO will be 0.92 mg, or 6 injections per treatment area (2 areas per treatment visit.
  Cohort B subjects will be given 1300 mg tranexamic acid PO TID prior to the day of the first and second CCH injections, the day of the first and second CCH injection, and the 3 days following the first and second CCH injections.
  Interventions: Drug: Collagenase Clostridium Histolyticum-Aaes; Drug: Lysteda 650 MG Oral Tablet
- Cohort C (Active Comparator): Per treatment area, subjects will be injected with up to 0.84 mg of QWO as 12 subcutaneous injections (0.3-mL injection administered as three 0.1-mL aliquots per injection), dependent on the amount of dimples (0.3 ml per dimple). A treatment area is defined as a left or right buttock, so patients may receive up to 1.84 mg, or 24 injections total (2 areas per treatment visit). The minimum dosage of QWO will be 0.92 mg, or 6 injections per treatment area (2 areas per treatment visit.
  Cohort C subjects will be given 1300 mg tranexamic acid PO TID prior to the day of the first, second, and third CCH injections, the day of the first, second, and third CCH injection, and the 3 days following the first, second, and third CCH injections.
  Interventions: Drug: Collagenase Clostridium Histolyticum-Aaes; Drug: Lysteda 650 MG Oral Tablet

INTERVENTIONS:
Drug: Collagenase Clostridium Histolyticum-Aaes — subjects will be injected with up to 0.84 mg of QWO as 12 subcutaneous injections (0.3-mL injection administered as three 0.1-mL aliquots per injection), dependent on the amount of dimples (0.3 ml per dimple).
  Other Names: QWO
Drug: Lysteda 650 MG Oral Tablet — Subjects will be given the therapeutic dose of tranexamic acid for menorrhagia, which is 1300 mg PO TID for up to 5 days during menstruation

SUMMARY:
This is an open-label, randomized, multiple dose IIR study to evaluate the effect of Lysteda™ on bruising following QWO™ injections to the buttocks in female subjects presenting with moderate to severe cellulite.

Following determination of eligibility based on inclusion/exclusion assessment, the subjects will be randomized to either Cohort A, Cohort B, or Cohort C, based on order of enrollment. Each Cohort will receive 3 Qwo™ treatments spaced 21 days apart, with 1300 mg of Lysteda™ TID PO at one, two, or all three treatments of Qwo™. Cohort A will be given tranexamic acid at the first treatment, Cohort B at the first and second treatment, and Cohort C at all three treatments. All buttock CCH injections will follow the on-label injection protocol.

Subjects will participate in the study for 65 days total, with an additional screening period of 14 days. There will be a total of 11 visits (Screening, Day 1, Day 4, Day 14, Day 22, Day 26, Day 36, Day 43, Day 47, Day 57, Day 65).

ELIGIBILITY:
Inclusion .

* Female > 18 and < 55 years of age.
* At the screening visit, have buttocks with moderate to severe cellulite based on the CR-PCSS.
* Be willing and able to comply with all protocol required visits and assessments.
* Be willing to apply sunscreen to the treatment areas before each exposure to the sun for the duration of the study.
* Is willing to refrain from exercise for 24 hours following each treatment.
* Be adequately informed and understand the nature and risks of the study.

Exclusion.

* Has a history of hypersensitivity or allergy to collagenase of any other excipient of CCH.
* At the screening visit, has none, almost none, or mild cellulite.
* At the screening visit, per the investigator, has cellulite that would require less than 6 injections per buttock, or more than 12 injections per buttock.
* Is pregnant and/or is breast-feeding or plans to become pregnant and/or to breast-feed during the course of the study, or 28 days after the last treatment.
* Is currently undergoing hormone replacement therapy or has undergone hormone replacement therapy in the past 6 months.
* Has a coagulation disorder which requires anticoagulant or antiplatelet medication during the study, or has taken anticoagulant or antiplatelet medication within 14 days before injections.
* Is currently taking oral contraceptive pills.
* Is currently a smoker, or has smoked within the last year prior to screening.
* Has a history of scarring due to keloids or abnormal wound healing.
* Has received previous treatment with CCH for cellulite, or any other cellulite treatment.
* Subject has any history of anemia or taking iron pills.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2022-04-22 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
Post CCH injection degree of bruising with TXA based on the Investigator Assessment of Bruising Severity Scale | 6 months
  Scale assessments completed at each follow-up visit. Bruising scale is 0-4, with 0 being no bruise and 4 being the worst bruise possible. A lower number on the bruising scales indicates a better outcome.
Post CCH injection degree of bruising with TXA based on Investigator Bruising Improvement Scale (I-BIS). | 6 months
  Scale assessments completed at each follow-up visit. Bruising scale is 0-4, with 0 being no bruise and 4 being the worst bruise possible. A lower number on the bruising scales indicates a better outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Luxurgery, New York, New York, United States